CLINICAL TRIAL: NCT03295123
Title: Outcome Children Born After Pregnancy Denial
Brief Title: Outcome of Children Born After Pregnancy Denial
Acronym: DENIGRO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: 2017-A00330-53
Record Dates: First submitted 2017-07-27; First posted 2017-09-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Child Development; Denial (Psychology); Disease; Personality Development
MeSH Terms: conditions — Rejection, Psychology; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone interview with the mother — it's a telephone survey about children's health

SUMMARY:
The objective of this study is to evaluate the impact of denial pregnancy on children's health ( anthropometric data, psychomotor development , disease) at different age of evaluation ( at birth, 9 months, 24 months and between 2 and 6 years post natal age).

The hypothesis is the denial of pregnancy may have repercussions on children's outcome.

ELIGIBILITY:
Inclusion Criteria:

* Child born after denial of pregnancy
* Child born at term ( > 37 weeks of gestation)
* Born between the 1st january 2009 and the 30th june 2015 at Maternité Regionale de Nancy

Exclusion Criteria:

* Mother's opposition
* Child doesn't' living in France

Ages: 1 Day to 8 Years | Sex: All
Age Groups: Child
Study Population: Every children born at term after denial of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
height (cm) | birth
  infants height will be recorded from their health booklet and compared to reference chart log
height (cm) | 9 months
  infants height will be recorded from their health booklet and compared to reference chart log
height (cm) | 24 months
  infants height will be recorded from their health booklet and compared to reference chart log
height (cm) | between 2 and 5 years
  infants height will be recorded from their health booklet and compared to reference chart log
weight (kg) | birth
  infants weight will be recorded from their health booklet and compared to reference chart log
weight (kg) | 9 months
  infants weight will be recorded from their health booklet and compared to reference chart log
weight (kg) | 24 months
  infants weight will be recorded from their health booklet and compared to reference chart log
weight (kg) | between 2 and 5 years
  infants weight will be recorded from their health booklet and compared to reference chart log

SECONDARY OUTCOMES:
psychomotor development | birth
  infants psychomotor development items will be recorded from their health booklet and compared to reference chart log
psychomotor development | 9 months
  infants psychomotor development items will be recorded from their health booklet and compared to reference chart log
psychomotor development | 24 months
  infants psychomotor development items will be recorded from their health booklet and compared to reference chart log
psychomotor development | between 2 and 5 years
  infants psychomotor development items will be recorded from their health booklet and compared to reference chart log
disease | birth
  all diseases which occured from birth will be recorded from their health booklet and compared to reference chart log
disease | 9 months
  all diseases which occured from birth will be recorded from their health booklet and compared to reference chart log
disease | 24 months
  all diseases which occured from birth will be recorded from their health booklet and compared to reference chart log
disease | between 2 and 5 years
  all diseases which occured from birth will be recorded from their health booklet and compared to reference chart log

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, France